CLINICAL TRIAL: NCT03912584
Title: Qualitative OCT Image Grading Study Comparing the P200TE and the P200TxE in Glaucoma Patients
Brief Title: Study Comparing the P200TE and the P200TxE in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT1038
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Results first posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Optical Coherence Tomographer (Other)
  Interventions: Device: P200TE; Device: P200TxE

INTERVENTIONS:
Device: P200TE — The P200TE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.
Device: P200TxE — The P200TxE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.

SUMMARY:
The study evaluates the image quality between two OCT devices.

DETAILED DESCRIPTION:
The objective of this study is to collect OCT scans to compare the qualitative B scan images produced by the P200TxE to the P200TE device in glaucoma subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 22 years of age or older who have full legal capacity to volunteer on the date the informed consent is signed;
* Subjects who can follow the instructions by the clinical staff at the clinical site,
* Subjects who agree to participate in the study;
* Subjects who have been diagnosed with glaucoma in the study eye as confirmed by the investigator;

Exclusion Criteria:

* Subjects unable to tolerate ophthalmic imaging;
* Subjects with ocular media not sufficiently clear to obtain acceptable OCT images;
* Subjects with any clinically significant ocular pathology except glaucoma, as determined by self-report and/or investigator assessment on the day of the study visit;
* Subjects who are not reliably tested with at least one Humphrey Field Analyzer (HFA) visual field (24-2 or 30-2, white on white) measured on the day of the study visit or within the previous year from the study visit, defined as fixation losses > 20% or false positives > 33%, or false negatives > 33%;
* Subjects with history of dementia or multiple sclerosis

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Ophthalmology Associates, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Optical Coherence Tomographer
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Optical Coherence Tomographer
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants] — Age 22 years or older, per inclusion criteria.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 5
    >=65 years | 5
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male or Female | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Glaucoma in Subject eye [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Qualitative B-Scan Assessment
Description: Scores will be based on a 4 point grading scale (0 to 3), with 0 corresponding to failure, 1 is poor, 2 is fair, and 3 is good.
  The four point scale is defined as follows:
  0 indicates the scan is a failure, and contains no clinically useful information. No relevant structures are visible in the scan.
  1. indicates the condition of the structure or feature being assessed is poor, and it contains very limited clinical utility.
  2. indicates the condition of the structure or feature being assessed is fair or average. It contains some useful clinical information and therefore provides adequate clinical utility.
  3. indicates the condition of the structure or feature being assessed is good. It contains useful clinical information. The clinical utility is high or good.
Time Frame: 1 day (start: April 29, 2019 - completed: April 30, 2019)
Population: The average score (0-3) for clinical utility and clinical quality for the P200TxE does not apply to P200TE scans, and the average score (0-3) for clinical utility and clinical quality for the P200TE does not apply to P200TxE scans. 10 subjects were imaged in total, however clinical utility and quality were measured separately for the three outcomes described below (1. Indy posterior scans, 2. Indy peripheral scans, 3. Monaco scans).
Measure: Mean (Standard Deviation); unit: Mean score on a scale (0-3)
Groups:
- Optical Coherence Tomographer - P200TE: P200TE: The P200TE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.
- Optical Coherence Tomographer - P200TxE: P200TxE: The P200TxE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.
Arm/Group | Optical Coherence Tomographer - P200TE | Optical Coherence Tomographer - P200TxE
Number analyzed (Participants) | 10 | 10
Mean score on a scale (0-3)
  Average score (0-3) for clinical utility and clinical quality Indy (P200TxE) Posterior scans: number analyzed (Participants) | 0 | 10
  Average score (0-3) for clinical utility and clinical quality Indy (P200TxE) Posterior scans |  | 2.78 (.45)
  Average score (0-3) for clinical utility and clinical quality Indy (P200TxE) Peripheral scans: number analyzed (Participants) | 0 | 10
  Average score (0-3) for clinical utility and clinical quality Indy (P200TxE) Peripheral scans |  | 2.77 (.46)
  Average score (0-3) for clinical utility and clinical quality Monaco (P200TE) scans: number analyzed (Participants) | 10 | 0
  Average score (0-3) for clinical utility and clinical quality Monaco (P200TE) scans | 2.08 (.64) |

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Analysis of safety will be assessed through adverse events reported by the site and documented on each subject's case report form. No AEs were recorded during this study.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Optical Coherence Tomographer P200TE: P200TE: The P200TE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.
Arm/Group | Optical Coherence Tomographer P200TE | Optical Coherence Tomographer - P200TxE
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Optical Coherence Tomographer: P200TE: P200TE: The P200TE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.
- Optical Coherence Tomographer: P200TxE: P200TxE: The P200TxE Ophthalmoscope provides widefield Scanning Laser Ophthalmoscope (SLO) fundus imaging and Optical Coherence Tomography (OCT) imaging in one device.
Arm/Group | Optical Coherence Tomographer: P200TE | Optical Coherence Tomographer: P200TxE
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT03912584/Prot_SAP_000.pdf